CLINICAL TRIAL: NCT06082076
Title: Dexmedetomidine Versus Ketamine to Prevent Shivering Associated With Intrathecal Anesthesia in Patients Undergoing Knee Arthroscopy:A Randomized, Controlled Double Blinded Study.
Brief Title: Prevention of Shivering Associated With Spinal Anesthesia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ahmed Galal Mohammed Mohammed, Mohammed Mohammed, Assiut University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Shivering and anesthesia
Record Dates: First submitted 2023-10-08; First posted 2023-10-13 (Actual); Last update posted 2023-10-13 (Actual); Status verified 2023-10

CONDITIONS: Shivering, Spinal Anesthesia
MeSH Terms: interventions — Dexmedetomidine; Ketamine; Meperidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group D (dexmedetomidine group) (Active Comparator)
  Interventions: Drug: Dexmedetomidine
- Group K (ketamine group) (Active Comparator)
  Interventions: Drug: Ketamine
- Group C (control group) (Placebo Comparator)
  Interventions: Drug: Meperidine

INTERVENTIONS:
Drug: Dexmedetomidine — Patients will receive dexmedetomidine 0.5 mcg/kg diluted in 10 mL of NS given as IV infusion over 10 min before induction of spinal anesthesia
  Arms: Group D (dexmedetomidine group)
Drug: Ketamine — Patient will will receive ketamine 0.5 mg/kg diluted in 10 mL of NS given as IV infusion over 10 min before induction of spinal anesthesia
  Arms: Group K (ketamine group)
Drug: Meperidine — If the tested drug hasn't stopped shivering patient will receive 0.25 mg/kg meperidine
  Arms: Group C (control group)

SUMMARY:
The aim of the study is to compare the effectiveness of prophylactic use of intravenous (IV) dexmedetomidine VS ketamine and meperidine(as a control group) in prevention of shivering associated with intrathecal anesthesia in patients undergoing knee arthroscopy

ELIGIBILITY:
Inclusion Criteria:

- BMI 20-30 Scheduled patients for knee arthroscopy under spinal anesthesia. American Society of Anesthesiologists (ASA) physical status: I and II

Exclusion Criteria:

* Patient refusal Aged less than 18 years or lesser than 150 cm in height Pregnant woman Allergy to the studied drugs. Patients with contraindications to spinal anesthesia. Patients with advanced decompensated cardiac, respiratory,renal or hepatic diseases, ASA III-IV Coagulopathy or thrombocytopenia CNS diseases as epilepsy, stroke or psychiatric illness.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Estimated)
Dates: Start 2023-11 (Estimated); Primary Completion 2024-11 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of shivering | During operation time
  Incidence of shivering post intrathecal anesthesia is recorded

CONTACTS AND LOCATIONS:
Overall Officials: Essam Ez Abdelhakeem, Professor, Study Director — Assiut University; Seham Mo Moeen, Professor, Study Director — Assiut University